CLINICAL TRIAL: NCT02991144
Title: A Phase 1/2, Open-Label Safety and Dose-Finding Study of Adeno-Associated Virus (AAV) Serotype 8 (AAV8)-Mediated Gene Transfer of Human Ornithine Transcarbamylase (OTC) in Adults With Late-Onset OTC Deficiency
Brief Title: Safety and Dose-Finding Study of DTX301 (scAAV8OTC) in Adults With Late-Onset Ornithine Transcarbamylase (OTC) Deficiency
Acronym: CAPtivate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 301OTC01; 2016-001057-40 (EudraCT Number)
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Results first posted 2022-12-23 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Ornithine Transcarbamylase (OTC) Deficiency
Keywords: Gene Transfer; OTC Deficiency; Urea Cycle Disorder
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease; Urea Cycle Disorders, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: DTX301 2.0 × 10^12 GC/kg (Experimental): DTX301 (scAAV8OTC) 2.0 × 10^12 GC/kg will be administered as a single peripheral IV infusion. A reactive corticosteroid taper regimen will be administered to control transient vector-induced hepatic effects. Sodium acetate will be used as a tracer to measure the rate of ureagenesis.
  Interventions: Genetic: scAAV8OTC; Drug: Reactive Corticosteroid Taper Regimen
- Cohort 2: DTX301 6.0 × 10^12 GC/kg (Experimental): DTX301 (scAAV8OTC) 6.0 × 10^12 GC/kg will be administered as a single peripheral IV infusion. A reactive corticosteroid taper regimen will be administered to control transient vector-induced hepatic effects. Sodium acetate will be used as a tracer to measure the rate of ureagenesis.
  Interventions: Genetic: scAAV8OTC; Drug: Reactive Corticosteroid Taper Regimen
- Cohort 3: DTX301 1.0 × 10^13 GC/kg (Experimental): DTX301 (scAAV8OTC) 1.0 × 10^13 GC/kg will be administered as a single peripheral IV infusion. A reactive corticosteroid taper regimen will be administered to control transient vector-induced hepatic effects. Sodium acetate will be used as a tracer to measure the rate of ureagenesis.
  Interventions: Genetic: scAAV8OTC; Drug: Reactive Corticosteroid Taper Regimen
- Cohort 4: DTX301 1.0x10^13 GC/kg + Prophylactic Corticosteroids (Experimental): A prophylactic corticosteroid taper regimen (oral prednisone [or prednisolone], 60 mg tapered over 9 weeks) will be administered before dosing with DTX301 (scAAV8OTC) to prevent or minimize transient vector-induced hepatic effects. DTX301 (scAAV8OTC) 1.0x10^13 GC/kg administered as a single peripheral IV infusion. Sodium acetate will be used as a tracer to measure the rate of ureagenesis.
  Interventions: Genetic: scAAV8OTC; Drug: Prophylactic Corticosteroid Taper Regimen

INTERVENTIONS:
Genetic: scAAV8OTC — non-replicating, recombinant scAAV8 encoding human ornithine transcarbamylase (OTC)
  Other Names: DTX301
Drug: Reactive Corticosteroid Taper Regimen — Oral prednisone [or oral prednisolone] 60 mg/day week 1, 40 mg/day Week 2, 30 mg/day Weeks 3 and 4, tapered by 5 mg/week Week 5 and beyond until liver enzymes return to baseline levels.
  Corticosteroid treatment will be considered when a participant's alanine aminotransferase (ALT) level exceeded the upper limit of normal (ULN) and the ALT increase was considered by the Investigator to be related to DTX301.
  Arms: Cohort 1: DTX301 2.0 × 10^12 GC/kg; Cohort 2: DTX301 6.0 × 10^12 GC/kg; Cohort 3: DTX301 1.0 × 10^13 GC/kg
Drug: Prophylactic Corticosteroid Taper Regimen — Oral prednisone [or oral prednisolone] 60 mg/day at least 5 days prior to DTX301 administration, tapered over 9 weeks.
  A prophylactic corticosteroid taper regimen will be administered to prevent or minimize transient vector-induced hepatic effects.
  Arms: Cohort 4: DTX301 1.0x10^13 GC/kg + Prophylactic Corticosteroids

SUMMARY:
This is a Phase 1/2, open-label, single arm, multicenter, safety and dose finding study of DTX301 in adults with late-onset OTC deficiency. The primary objective of the study is to determine the safety of single intravenous (IV) doses of DTX301.

DETAILED DESCRIPTION:
Eligible participants will receive a single IV infusion of DTX301. Dose escalation will be conducted according to a model that uses the collected data to predict the safety profile of the dose in order to determine the optimal biological dose (OBD). The decision to proceed to the next dose cohort will be made after the data monitoring committee (DMC) has evaluated the safety data for all participants in a dosing cohort. Participants will be followed for 52 weeks after dosing. After completion of this study, participants will be asked to enroll in a 4-year extension study to evaluate the long term (a total of 5 years) safety and efficacy of DTX301.

This study was previously posted by Dimension Therapeutics, which has been acquired by Ultragenyx.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females ≥18 years of age with documented diagnosis of late onset (defined as first manifestation of signs and symptoms at ≥1 month of age) OTC deficiency, confirmed via enzymatic, biochemical, or molecular testing
2. Documented history of ≥1 symptomatic hyperammonemia event with ammonia ≥100 µmol/L.
3. Subject's OTC deficiency is stable as evidenced by either a) no clinical symptoms of hyperammonemia OR b) an ammonia level <100 µmol/L within the 4 week period preceding the Screening visit.
4. On ongoing daily stable dose of ammonia scavenger therapy for ≥4 weeks.
5. Males and all females of childbearing potential must be willing to use effective contraception at the time of administration of gene transfer and for the 52 weeks following administration of DTX301

Key Exclusion Criteria:

1. At Screening or Baseline (Day 0), plasma ammonia level ≥ 100 μmol/L for patients who historically maintain normal ammonia levels; OR plasma ammonia level ≥ 200 μmol/L for patients who historically are not able to fully control ammonia levels with baseline management; OR signs and symptoms of hyperammonemia.
2. Liver transplant, including hepatocyte cell therapy/transplant.
3. History of liver disease
4. Significant hepatic inflammation or cirrhosis
5. Serum creatinine >2.0 mg/dL.
6. Participation in another investigational medicine study (including another gene transfer trial) within 3 months of Screening
7. Pregnant or nursing

Note additional inclusion/exclusion criteria may apply, per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (9):
- United States (4):
  - The Children's Hospital Colorado, Aurora, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University Hospital Cleveland Medical Center/Case Western Reserve University, Cleveland, Ohio
- Alberta's Children's Hospital, Calgary, Alberta, Canada
- Spain (2):
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruna
  - Hospital Universitario de Cruzes, Barakaldo, Vizcaya
- United Kingdom (2):
  - National Hospital for Neurology & Neurosurgery, London, London City
  - Queen Elizabeth Hospital, Birmingham

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 27 subjects were screened for the study, 16 of whom were enrolled. Of the 16 participants enrolled, 5 participants discontinued the study before receiving DTX301, and were not assigned to a treatment arm.
Groups:
- Cohort 1: DTX301 2.0 × 10^12 GC/kg: DTX301 (scAAV8OTC) 2.0 × 10^12 GC/kg administered as a single peripheral intravenous (IV) infusion.
- Cohort 2: DTX301 6.0 × 10^12 GC/kg: DTX301 (scAAV8OTC) 6.0 × 10^12 GC/kg administered as a single peripheral IV infusion.
- Cohort 3: DTX301 1.0 × 10^13 GC/kg: DTX301 (scAAV8OTC) 1.0 × 10^13 GC/kg administered as a single peripheral IV infusion.
- Cohort 4: DTX301 1.0x10^13 GC/kg + Prophylactic Corticosteroids: Oral prednisone (or prednisolone), 60 mg tapered over 9 weeks, initiated before dosing with DTX301 (scAAV8OTC) and administered through Week 4. DTX301 (scAAV8OTC) 1.0x10^13 GC/kg administered as a single peripheral IV infusion.
Period: Overall Study
Arm/Group | Cohort 1: DTX301 2.0 × 10^12 GC/kg | Cohort 2: DTX301 6.0 × 10^12 GC/kg | Cohort 3: DTX301 1.0 × 10^13 GC/kg | Cohort 4: DTX301 1.0x10^13 GC/kg + Prophylactic Corticosteroids
Started | 3 | 3 | 3 | 2
Completed | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: DTX301 2.0 × 10^12 GC/kg: DTX301 (scAAV8OTC) 2.0 × 10^12 GC/kg administered as a single peripheral IV infusion.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: DTX301 2.0 × 10^12 GC/kg | Cohort 2: DTX301 6.0 × 10^12 GC/kg | Cohort 3: DTX301 1.0 × 10^13 GC/kg | Cohort 4: DTX301 1.0x10^13 GC/kg + Prophylactic Corticosteroids | Total
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (11.06) | 27.7 (1.15) | 26.7 (7.09) | 30.5 (13.44) | 29.2 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 7
  Male | 2 | 1 | 1 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 2 | 3 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 3 | 3 | 2 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Rate of Ureagenesis [Mean (Standard Deviation); unit: μmol*h/kg] — Rate of ureagenesis (as measured by the generation of [13C]urea over 4 hours; see outcome measure 2 for details). Baseline is defined as the average of all non-missing assessments taken before the study drug administration. If the absolute difference of results between Screening and Day 1 was ≥ 25% of normal rate of ureagenesis, then the screening value is defined as the baseline.
  μmol*h/kg | 166.293 (28.0167) | 103.329 (76.9798) | 115.492 (71.0753) | 174.678 (210.9140) | 136.791 (88.4373)
Area Under the Curve From Time Zero to 24 Hours (AUC0 24) of Plasma Ammonia [Mean (Standard Deviation); unit: μmol*h/L] — Baseline is defined as the Day -1 result. Population: participants with a baseline assessment
  μmol*h/L
    number analyzed (Participants) | 3 | 3 | 1 | 2 | 9
    (all) | 1831.78 (1445.240) | 2153.74 (1406.173) | 4444.76 (NA) — 1 participant analyzed | 1834.39 (1091.019) | 2230.01 (1370.847)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Deaths, and TEAEs Leading to Discontinuation
Description: AE: any untoward medical occurrence regardless of its causal relationship to study product. TEAE: any event not present before exposure to study product or any event already present that worsens in either intensity or frequency after exposure to study product. SAE: any event that results in death; is immediately life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; is an important medical event, according to the investigator. AE intensity was rated as Grade 1 (mild), 2 (moderate), 3 (severe), 4 (life threatening), or 5 (death) according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE). The relationship or association of the study product in causing or contributing to the AE was characterized as: unrelated; possible; probably; definite.
Time Frame: AEs Prior to Dosing: From signing the informed consent form (ICF) to first dose of study drug. TEAEs: From first dose of study drug up to End of Study (Week 52).
Population: Safety Set: all participants who received DTX301.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DTX301 2.0 × 10^12 GC/kg | Cohort 2: DTX301 6.0 × 10^12 GC/kg | Cohort 3: DTX301 1.0 × 10^13 GC/kg | Cohort 4: DTX301 1.0x10^13 GC/kg + Prophylactic Corticosteroids
Number analyzed (Participants) | 3 | 3 | 3 | 2
Participants
  Any AE prior to dosing | 1 | 1 | 0 | 1
  Any TEAE | 3 | 3 | 3 | 2
  Any serious TEAE | 0 | 0 | 0 | 1
  Any TEAE with grade >=3 | 0 | 0 | 0 | 1
  Any study drug-related TEAE | 2 | 1 | 3 | 2
  Any TEAE related to corticosteroid regimen | 1 | 0 | 1 | 1
  Any hyperammonemic crisis-related TEAE | 0 | 0 | 0 | 1
  Any study drug-related serious TEAE | 0 | 0 | 0 | 0
  Any study drug-related TEAE with grade >=3 | 0 | 0 | 0 | 0
  Any TEAE leading to study discontinuation | 0 | 0 | 0 | 0
  Any adverse event leading to death | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline Over Time in Rate of Ureagenesis
Description: The change from baseline in the rate of ureagenesis (as measured by the generation of [13C]urea over 4 hours) as determined by gas chromatography mass spectrometry over time to 52 weeks after the IV administration of DTX301. Sodium acetate was used as a tracer to measure the rate of ureagenesis.
  Rate of ureagenesis was derived in the following manner:
  1. Derive area under the curve from time zero to 240 minutes (AUC0-240min) of absolute 13C-urea (µmol/l/min) estimated by the linear trapezoidal rule
  2. Derive percent of normal AUC0-240min of absolute 13C-urea by dividing AUC0-240min of absolute 13C-urea (µmol*min/L) by 669.56 µmol*min/L (i.e. the AUC0-240min of absolute 13C-urea for an adult control)
  3. Derive rate of ureagenesis by multiplying % of normal AUC0-240min of absolute 13C-urea by 300 µmol*h/kg (i.e. the approximate rate of ureagenesis in healthy adults).
Time Frame: Baseline (Day 0), Weeks 6, 12, 20, 24, End of Study (Week 52). AUC was derived based on the following time points: 0.5, 1, 1.5, 2, 3, and 4 hours postdose.
Population: Safety Set: all participants who received DTX301.
Measure: Mean (Standard Deviation); unit: μmol*h/kg
Arm/Group | Cohort 1: DTX301 2.0 × 10^12 GC/kg | Cohort 2: DTX301 6.0 × 10^12 GC/kg | Cohort 3: DTX301 1.0 × 10^13 GC/kg | Cohort 4: DTX301 1.0x10^13 GC/kg + Prophylactic Corticosteroids
Number analyzed (Participants) | 3 | 3 | 3 | 2
μmol*h/kg
  Change at Week 6 | 41.139 (83.3604) | 46.857 (105.9147) | -29.017 (127.2471) | 14.586 (17.3499)
  Change at Week 12 | 2.363 (51.2516) | 20.897 (56.9733) | 7.544 (133.1715) | 65.781 (33.9137)
  Change at Week 20 | 32.929 (71.0500) | 77.465 (67.1567) | -0.194 (112.5922) | 67.103 (102.5409)
  Change at Week 24 | 42.540 (136.5861) | 65.513 (50.5169) | 45.114 (147.5760) | 63.854 (106.7694)
  Change at End of Study (Week 52) | 109.611 (171.0689) | 114.446 (98.8701) | 10.016 (47.9128) | 128.023 (131.6469)

3. Secondary Outcome: Change From Baseline Over Time in Area Under the Curve From Time Zero to 24 Hours (AUC0-24) of Plasma Ammonia
Time Frame: Baseline (Day 0), Weeks 6, 12, 24, End of Study (Week 52). AUC was derived based on predose (time 0) and approximately 2, 4, 8, 12, 16, 20, 24 hours (±5 minutes) postdose.
Population: Safety Set: all participants who received DTX301. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: μmol*h/L
Arm/Group | Cohort 1: DTX301 2.0 × 10^12 GC/kg | Cohort 2: DTX301 6.0 × 10^12 GC/kg | Cohort 3: DTX301 1.0 × 10^13 GC/kg | Cohort 4: DTX301 1.0x10^13 GC/kg + Prophylactic Corticosteroids
Number analyzed (Participants) | 3 | 3 | 3 | 2
μmol*h/L
  Change at Week 6: number analyzed (Participants) | 2 | 3 | 1 | 2
  Change at Week 6 | 97.69 (104.381) | -1334.27 (1271.205) | -3790.83 (NA) — 1 participant analyzed | -1095.20 (785.719)
  Change at Week 12: number analyzed (Participants) | 3 | 3 | 1 | 2
  Change at Week 12 | -264.07 (1471.172) | -1384.95 (1279.839) | -3827.36 (NA) — 1 participant analyzed | -1242.69 (931.242)
  Change at Week 24: number analyzed (Participants) | 3 | 3 | 1 | 2
  Change at Week 24 | -252.54 (586.131) | -1065.48 (1024.167) | -3978.51 (NA) — 1 participant analyzed | -1276.25 (943.999)
  Change at End of Study (Week 52): number analyzed (Participants) | 3 | 2 | 1 | 2
  Change at End of Study (Week 52) | -381.54 (1116.898) | -387.02 (277.086) | -594.76 (NA) — 1 participant analyzed | -359.17 (1641.519)

ADVERSE EVENTS:
Time Frame: All Cause Mortality: from screening up to End of Study (Week 52). Adverse Events and Serious Adverse Events: From first dose of study drug up to End of Study (Week 52).
Description: 2 enrolled participants died before receiving DTX301, and were not assigned to a treatment arm. These participants are reflected in the 'total' column of the all-cause mortality table.
Groups:
- DTX301 2.0 × 10^12 GC/kg: DTX301 (scAAV8OTC) 2.0 × 10^12 GC/kg administered as a single peripheral IV infusion.
- DTX301 6.0 × 10^12 GC/kg: DTX301 (scAAV8OTC) 6.0 × 10^12 GC/kg administered as a single peripheral IV infusion.
- DTX301 1.0 × 10^13 GC/kg: DTX301 (scAAV8OTC) 1.0 × 10^13 GC/kg administered as a single peripheral IV infusion.
- DTX301 1.0x10^13 GC/kg + Prophylactic Corticosteroids: Oral prednisone (or prednisolone), 60 mg tapered over 9 weeks, initiated before dosing with DTX301 (scAAV8OTC) and administered through Week 4. DTX301 (scAAV8OTC) 1.0x10^13 GC/kg administered as a single peripheral IV infusion.
- Total: All Participants
Arm/Group | DTX301 2.0 × 10^12 GC/kg | DTX301 6.0 × 10^12 GC/kg | DTX301 1.0 × 10^13 GC/kg | DTX301 1.0x10^13 GC/kg + Prophylactic Corticosteroids | Total
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/2 | 2/16
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 1/2 | 1/11
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 2/2 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTX301 2.0 × 10^12 GC/kg (N=3) | DTX301 6.0 × 10^12 GC/kg (N=3) | DTX301 1.0 × 10^13 GC/kg (N=3) | DTX301 1.0x10^13 GC/kg + Prophylactic Corticosteroids (N=2) | Total (N=11)
Hyperammonaemic Crisis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 — There were 2 serious adverse events of hyperammonaemic crisis that occurred in 1 subject post-dosing.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTX301 2.0 × 10^12 GC/kg (N=3) | DTX301 6.0 × 10^12 GC/kg (N=3) | DTX301 1.0 × 10^13 GC/kg (N=3) | DTX301 1.0x10^13 GC/kg + Prophylactic Corticosteroids (N=2) | Total (N=11)
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Cushingoid (Endocrine disorders) | 1 | 0 | 1 | 0 | 2
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2
Catheter Site Pain (General disorders) | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 2
Feeling Abnormal (General disorders) | 0 | 0 | 1 | 1 | 2
Feeling Jittery (General disorders) | 0 | 0 | 0 | 1 | 1
Gait Disturbance (General disorders) | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1
Gallbladder Polyp (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 2
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Exposure To Sars-Cov-2 (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 1 | 0 | 2
Liver Function Test Abnormal (Investigations) | 0 | 0 | 1 | 0 | 1
Liver Function Test Increased (Investigations) | 0 | 0 | 0 | 2 | 2
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 2 | 2 | 5
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Neuropathy Peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1 | 2
Aggression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Claustrophobia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 2
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Phonophobia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT02991144/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT02991144/SAP_001.pdf